CLINICAL TRIAL: NCT04495803
Title: Augmented Cognitive Behavioural Group Therapy for Perinatal Anxiety During a Global Pandemic (COVID-19)
Brief Title: Augmented CBGT for Perinatal Anxiety During a Global Pandemic (COVID-19)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: St. Joseph's Healthcare Hamilton (Other)
Responsible Party: Principal Investigator, Sheryl Green, Clinical Health Psychologist, St. Joseph's Healthcare Hamilton
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CBT-COVID
Record Dates: First submitted 2020-07-30; First posted 2020-08-03 (Actual); Last update posted 2022-05-04 (Actual); Status verified 2022-05

CONDITIONS: Perinatal Anxiety; Covid19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental (Experimental): After an initial assessment to confirm eligibility, the experimental group will receive 8 weekly sessions (2 hours long) of our augmented group CBT for perinatal anxiety during a global pandemic (n=6 per group). Participants will be re-assessed at post-treatment and at a 3-month follow-up to determine the effectiveness of the treatment and whether these effects are maintained in the long-term.
  Interventions: Other: Cognitive Behavioural Group Therapy for Perinatal Anxiety

INTERVENTIONS:
Other: Cognitive Behavioural Group Therapy for Perinatal Anxiety — The treatment consists of cognitive and behavioural strategies for treating anxiety, tailored specifically to a perinatal/postpartum population. Additional strategies for COVID-19 specific worry content have been included.

SUMMARY:
This study will evaluate the effectiveness of an augmented version of our current evidence-based Cognitive Behavioural Group Therapy (CBGT) for perinatal anxiety protocol with cognitive and behavioural strategies composed of critical COVID-related anxiety, worry, and impact content.

ELIGIBILITY:
Inclusion Criteria:

* Females, aged 18-45 years
* Pregnant or up to six months postpartum
* Primary diagnosis of an anxiety disorder, as per the MINI for DSM-5, with or without comorbid depression
* No concurrent psychological treatment
* Not taking psychoactive medication or medication is stable in dose and type for at least 8 weeks prior to the study (as per Canadian Psychiatric Guidelines) and throughout study duration (participants will not be excluded from treatment if medication/dose changes during the study duration, however, they must notify the study team immediately)
* Fluent in English in order to understand the consent and group material

Exclusion Criteria:

* Severe depression/suicidality
* Primary diagnosis other than an anxiety disorder
* Psychotic or current substance/alcohol use disorder

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 68 (Actual)
Dates: Start 2020-09-01 (Actual); Primary Completion 2021-09-01 (Actual); Study Completion 2021-09-01 (Actual)

PRIMARY OUTCOMES:
State-Trait Inventory of Cognitive and Somatic Anxiety (STICSA) | 8 weeks
  Changes in anxiety symptoms will be assessed through the STICSA to examine whether our augmented CBT for perinatal anxiety during a global pandemic is effective in reducing anxiety symptoms. Items on the STICSA are rated on a 4-point likert scale ranging from 1 (not at all) to 4 (very much so), with higher scores indicating worse anxiety symptoms. The STICSA has two subscales (i.e., cognitive subscale and somatic subscale) and a total score that will be used in analysis. Ten items comprise the cognitive subscale, meaning scores can range from 10-40. Eleven items comprise the somatic subscale, meaning scores can range from 11 -44. The total score is a sum of both subscales with possible total scores in the range of 21-84.

SECONDARY OUTCOMES:
Intolerance of Uncertainty Scale (IUS) | 8 weeks
  Due to the level of ongoing uncertainty that exists surrounding COVID-19, changes in intolerance of uncertainty will be assessed by the 27-item IUS to examine whether our augmented CBT for perinatal anxiety during a global pandemic is effective in reducing intolerance of uncertainty. The IUS can be scored across two-factors, in addition to a total score. Factor 1 includes items assessing uncertainty as having negative behavioural and self-referent implications (e.g., uncertainty keeps me from living a full life) and Factor 2 assesses uncertainty as being unfair and spoiling things in life (e.g., I can't stand being taken by surprise). Items are rated on a 5-point Likert type scale ranging from 1 (not at all characteristic of me) to 5 (entirely characteristic of me).
Penn State Worry Questionnaire (PSWQ) | 8 weeks
  Changes in worry symptoms will be assessed by the PSWQ. The PSWQ is a 16-item self-administered tool designed to assess worry symptoms. Items are assessed on a 5-point Likert scale ranging from 1 (not at all typical of me) to 5 (very typical of me), with higher scores indicating increased worry.
Edinburgh Postnatal Depression Scale (EPDS) | 8 weeks
  Changes in mood symptoms will be assessed through the EPDS. Items on the EPDS are rated from 0-3, with higher total scores indicating more depressive symptoms. Possible scores on the EPDS range from 0-30. A clinical cut-off of 13 is used to indicate probable depression.
COVID-19 Stress Scales (CSS) | 8 weeks
  Changes in worry and anxiety associated with COVID-19 will be examined using the CSS. The CSS is a 36-item self-report scale designed to measure worry and anxiety associated with the novel COVID-19 pandemic. Each item is rated on a 5-point Likert scale ranging from 0 to 4. The CSS has 5 subscales: danger and contamination fears, fears about economic consequences, xenophobia, compulsive checking and traumatic stress symptoms.
Pregnancy-Related Anxiety Questionnaire-Revised (PRAQ-R2) | 8 weeks
  Changes in pregnancy-specific anxiety will be assessed with the PRAQ-R2. Items are scored on 5-point Likert scale. Respondents are asked to circle the answer that applies most accurately to their situation and higher scores are reflective of greater pregnancy-specific anxiety. The PRAQ-R2 contains three subscales: fear of giving birth, worries about bearing a handicapped child, and concern about own appearance.
Postpartum Specific Anxiety Scale (PSAS) | 8 weeks
  Changes in postpartum-specific anxiety will be assessed with the PSAS. Items are scored on a 4-point Likert scale (0-3), with higher scores indicating greater anxiety symptoms. The PSAS has 4 subscales: maternal competence and attachment, infant safety and welfare, practical infant care, and psychosocial adjustment to motherhood.
Overall Anxiety Severity and Impairment Scale (OASIS) | 8 weeks
  Changes in severity and impairment associated with anxiety will be assessed with the OASIS. Respondents are asked to circle that answer that best describes their experience over the past week and items are scored on a 5-point Likert scale.
Parenting Sense of Competence Scale (PSOC) | 8 weeks
  Changes in parenting self-efficacy will be assessed with the PSOC. The PSOC is a 17-item self-report scale, in which items are scored on a 6-point Likert scale ranging from 1 (strongly disagree) to 6 (strongly agree), with higher scores reflecting greater parenting sense of competency.
Abbreviated Dyadic Adjustment Scale (ADAS) | 8 weeks
  Changes in relationship satisfaction and adjustment will be assessed with the ADAS. The ADAS is a 7-item self-report scale, in which six of the items are scored on a 6-point Likert Scale, with higher scores reflecting greater relationship satisfaction. Item seven provides a global 'overall happiness' rating and is scored on 7-point Likert Scale ranging from 0 (extremely unhappy) to 6 (perfect).
Social Provisions Scale (SPS) | 8 weeks
  Changes in perceived social support will be assessed with the SPS. Items are scored on a 4-point Likert scale ranging from 1 (strongly disagree) to 4 (strongly agree), with higher scores indicating higher levels of perceived social support. The SPS has 6 subscales assessing dimensions of attachment, social integration, reassurance of worth, guidance, nurturance and reliance.
Maternal Antenatal Attachment Scale (MAAS) | 8 weeks
  Changed in maternal attachment and bonding to the fetus will be assessed with the MAAS. For each item, respondents are asked to indicate the frequency in which each experience has occurred within the previous two weeks. The MAAS has two subscales that assess dimensions of quality of attachment and intensity of preoccupation. Items are scored on a 5-point Likert scale and scores range from 19 to 95 with higher scores indicating a higher level of attachment to the fetus.
Postpartum Bonding Questionnaire (PBQ) | 8 weeks
  Changes in maternal bonding with the infant will be assessed with the PBQ. Items are scored on a 6-point Likert scale ranging from 0 (always) to 5 (never), with higher scores indicating lower levels of bonding with the infant. The PBQ has four subscales: general bonding, rejection and pathological anger, anxiety about the infant, and incipient abuse.
Client Satisfaction Questionnaire (CSQ) | 8 weeks
  Client satisfaction of the augmented CBT for perinatal anxiety during a global pandemic will be assessed with the CSQ. Items are scored on a 4-point Likert scale from 1 to 4, with higher scores indicating higher levels of satisfaction with services.
Perceived Stress Scale (PSS) | 8 weeks
  Changes in participants perceived level of stress will be assessed with the PSS. The PSS is a 14-item self-report scale, with items scored on a 5-point Likert scale from 0 to 4, with higher total scores indicating higher perceived stress.

CONTACTS AND LOCATIONS:
Locations (1):
- St. Joseph's Healthcare Hamilton, Hamilton, Ontario, Canada